CLINICAL TRIAL: NCT00609323
Title: A Randomized, Double-Blind, Crossover Study Comparing Pliaglis™ (Lidocaine and Tetracaine) Cream 7%/7% to Placebo Cream When Applied for 60 Minutes in the Treatment of Patients With Postherpetic Neuralgia
Brief Title: Lidocaine and Tetracaine Cream to Treat Postherpetic Neuralgia (PHN)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ZARS Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SCP-403
Record Dates: First submitted 2008-01-18; First posted 2008-02-07 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-03

CONDITIONS: Postherpetic Neuralgia
Keywords: Pain; postherpetic neuralgia
MeSH Terms: conditions — Neuralgia, Postherpetic; Pain | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: lidocaine and tetracaine cream 7%/7%
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: lidocaine and tetracaine cream 7%/7% — One treatment of up to 400 cm2 Cream applied for 60 minutes.
  Other Names: Pliaglis™
  Arms: 1
Drug: Placebo — One treatment of up to 400 cm2 Cream applied for 60 minutes.
  Arms: 2

SUMMARY:
Pliaglis™ (lidocaine and tetracaine) Cream 7%/7% is a topical local anesthetic cream that forms a pliable peel on the skin when exposed to air. When applied to intact skin, Pliaglis provides local dermal analgesia by the release of lidocaine and tetracaine from the peel into the skin.

Pliaglis is currently approved in the United States for use on intact skin in adults to provide topical local analgesia for superficial dermatological procedures such as dermal filler injection, pulsed dye laser therapy, and facial laser resurfacing.

This study will evaluate lidocaine and tetracaine cream 7%/7% for the treatment of pain associated with postherpetic neuralgia (PHN).

DETAILED DESCRIPTION:
The objectives of the study are 1) to compare the clinical efficacy of lidocaine and tetracaine cream 7%/7% with placebo cream in the treatment of neuropathic pain associated with postherpetic neuralgia (PHN) and 2) to monitor the nature and frequency of adverse events following a single, 60-minute application of lidocaine and tetracaine cream 7%/7% and placebo cream.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of PHN.
* Painful PHN areas not located on the face, eye, or in the hair.
* At least 3 months post-vesicle crusting.

Exclusion Criteria:

* Has broken skin at the target treatment site.
* Is currently on certain prescription medications.
* Doesn't meet criteria due to physical exam findings or medical history.
* Female that is pregnant, breastfeeding, or of childbearing potential and not practicing adequate birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-01; Primary Completion 2008-07 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Pain will be rated using the Numeric Pain Rating Scale (NPRS). Patients will rate: Worst pain over the last 24 hours, Least pain over the last 24 hours, Average pain over the last 24 hours, Present pain intensity. | 24 hours after treatment
Area of allodynia will be mapped at baseline and at the treatment sessions. | 1-2 weeks between study treatments
Intensity of allodynia | Baseline, 4 hours, 9 hours, 24 hours after treatment
Patient global impression of change. | 9 & 24 hours after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — ZARS Pharma
Locations (6):
- United States (6):
  - ZARS Pharma Clinical Site, Lexington, Kentucky
  - ZARS Pharma Clinical Site. Reference: SCP-403, High Point, North Carolina
  - ZARS Pharma Clinical Site. Reference: SCP-403, Winston-Salem, North Carolina
  - ZARS Pharma Clinical Site, Norman, Oklahoma
  - ZARS Pharma Clinical Site, Oklahoma City, Oklahoma
  - ZARS Pharma Clinical Site, San Antonio, Texas